CLINICAL TRIAL: NCT03848559
Title: Airway Management With Simulated Microgravity Using a Submerged Model
Acronym: AirMicroMod
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: AirMicroMod
Record Dates: First submitted 2019-02-14; First posted 2019-02-20 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Airway Management; Emergency Medicine
MeSH Terms: interventions — Airway Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Airway device placement (Experimental): airway device is placed during the dive
  Interventions: Device: Airway management with a submerged model

INTERVENTIONS:
Device: Airway management with a submerged model — Airway management with a submerged manikin using different airway devices in randomized order

SUMMARY:
Trained anesthesiologist- or emergency physician-divers will perform an airway management in simulated microgravity on a submerged model.

DETAILED DESCRIPTION:
Trained anesthesiologist- or emergency physician-divers participate in the study. Simulated microgravity during spaceflight is obtained by using a submerged model. Full-torso manikins is going to be used for performing airway management. Each diver attempted airway management with each device (laryngeal mask, laryngeal tube, orotracheal intubation with video-assisted laryngoscope. The time for airway protection will be measured as well as the success rate.

ELIGIBILITY:
Inclusion Criteria:

* Anaesthesiologist with diver licence or Emergency physician with diver license

Exclusion Criteria:

* All other

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Number of inserts | after 5 minutes
  Summarizing the number of Intubation attempts or attempts to place the supraglottic airway
Time to first ventilation | after 5 minutes
  Time from beginning with the airway manoeuvre (taking the decice) until successful airway secure and first ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Hinkelbein, MD, PhD, Study Chair — UK Köln
Locations (1):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided